CLINICAL TRIAL: NCT01049308
Title: Cognitive Impairment as a Risk for the Admission-Readmission Cycle Seen in Veterans With Heart Failure: Closing the Adherence Gap
Brief Title: Cognitive Problems in Veterans With Heart Failure
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: RRP 09-166
Record Dates: First submitted 2010-01-12; First posted 2010-01-14 (Estimated); Results first posted 2014-11-24 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2014-08

CONDITIONS: Heart Failure; Cognition Disorders
Keywords: heart failure; cognitive disorders; medication adherence; patient readmissions
MeSH Terms: conditions — Heart Failure; Cognition Disorders; Cognitive Dysfunction; Medication Adherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Heart Failure: veteran population with documented heart failure

SUMMARY:
We assessed the prevalence of cognitive/memory problems in veteran patients with heart failure, and evaluated its relationship to medication compliance.

DETAILED DESCRIPTION:
Heart failure (HF) is a costly, chronic, and complex condition that impacts veterans' quality of life, morbidity, and mortality. In the VA population up to 20% of patients are readmitted for HF within 30 days. Non-adherence to prescribed medication and self-care regimens in patients with HF is known to lead to increased morbidity, including readmissions. Cognitive impairment (CI) has been shown to predict nonadherence in elderly people without HF, however, this link has not been studied in HF populations. In the non-veteran population, HF patients are known to have an increased prevalence of cognitive impairment (CI), however, no existing study has determined the extent and type of CI in veterans with HF.

This pilot study was designed as a descriptive cross-sectional study as a pre-implementation effort with following goals: (1) determine the prevalence of CI in veterans with all-cause HF in an outpatient setting; (2) quantitatively describe the extent of CI in this population; (3) qualitatively describe neuropsychological domains affected by CI; (4) evaluate the association of CI with medication adherence and other clinical variables.

All consenting eligible outpatients in our VA HF clinic underwent a simple screening test for CI (Saint Louis University Mental Status Exam). Demographic and clinical variables were collected by patient interviews and chartg reviews, and included Geriatric Depression Scale and questionnaires about medication-taking behaviors. All subjects were invited back for 30-day direct pill count of all their routinely prescribed medications. Subjects who screened positive for CI were invited back for a modified battery of neuropsychological tests to determine the cognitive domains affected. Subjects will also be followed after the 12-month study period to collect data on hospital readmissions.

ELIGIBILITY:
Inclusion Criteria:

* Patients with established diagnosis of clinical heart failure
* English-speaking
* Able to provide informed consent
* Able to participate in cognitive function testing
* Age over 18

Exclusion Criteria:

* Life expectancy < 6 months
* Documented dementia requiring a caregiver

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: veteran patients enrolled in outpatient heart failure clinic
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2010-02; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helme Silvet, MD, Principal Investigator — VA Loma Linda Healthcare System, Loma Linda, CA
Locations (1):
- VA Loma Linda Healthcare System, Loma Linda, CA, Loma Linda, California, United States

REFERENCES:
- [Result] Hawkins LA, Kilian S, Firek A, Kashner TM, Firek CJ, Silvet H. Cognitive impairment and medication adherence in outpatients with heart failure. Heart Lung. 2012 Nov-Dec;41(6):572-82. doi: 10.1016/j.hrtlng.2012.06.001. Epub 2012 Jul 10. PMID 22784869

RESULTS

PARTICIPANT FLOW:
Period: Evaluation of Cognitive Impairment
Arm/Group | Heart Failure
Started | 251
Completed | 251
Not Completed | 0
Period: Pill Counts
Arm/Group | Heart Failure
Started | 251
Completed | 168
Not Completed | 83
Not completed — Withdrawal by Subject | 83

BASELINE CHARACTERISTICS:
Groups:
- Group 1: veteran population with documented heart failure
Arm/Group | Group 1
Number analyzed (Participants) | 251
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.4 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 247
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 34
  White | 180
  More than one race | 0
  Unknown or Not Reported | 37
Living arrangement [Number; unit: participants]
  Live alone | 68
  Live with spouse/partner | 142
  Live with children | 17
  Other | 22
  Not reported | 2
education [Number; unit: participants]
  Less than high school | 25
  High school diploma | 60
  Some college | 103
  College degree or above | 60
  Not reported/unknown | 3
self-perceived financial status [Number; unit: participants]
  Does not affect ability to care for health | 111
  Affects ability to care for health | 110
  Not reported/unknown | 30
Diabetes (I or II) [Number; unit: participants]
  Have diagnosis | 134
  Do not have diagnosis | 117
Coronary Artery Disease [Number; unit: participants]
  Have diagnosis | 160
  Do not have diagnosis | 91
Hypertension [Number; unit: participants]
  Have diagnosis | 193
  Do not have diagnosis | 58
Obstructive sleep apnea [Number; unit: participants]
  Have diagnosis | 68
  Do not have diagnosis | 183
History of atrial fibrillation [Number; unit: participants]
  Yes | 82
  No | 169
History of stroke [Number; unit: participants]
  Yes | 26
  No | 225
Systolic blood pressure [Mean (Standard Deviation); unit: mm hG] | 125.8 (19.67)
Thiamine level [Mean (Standard Deviation); unit: nmol/L] | 169 (95.60)
Vitamin B12 level [Mean (Standard Deviation); unit: pg/mL] | 556.8 (298.26)
Hemoglobin level [Mean (Standard Deviation); unit: g/dL] | 13.6 (2.19)
Serum creatinine level [Mean (Standard Deviation); unit: mg/dL] | 1.59 (1.84)
Thyroid-stimulating hormone [Mean (Standard Deviation); unit: uiU/mL] | 2.99 (4.39)
Brain natriuretic peptide level [Mean (Standard Deviation); unit: pg/mL] | 274.7 (497)
Hemoglobin A1c [Mean (Standard Deviation); unit: %] | 6.8 (1.5)
Heart Failure duration [Number; unit: participants]
  Less than 1 year | 22
  1-5 years | 104
  Greater than 5 years | 123
  Not reported/unknown | 2
Heart failure cause [Number; unit: participants]
  Ischemic | 131
  Non-ischemic | 107
  Not reported/unknown | 13
Left ventricular ejection fraction [Number; unit: participants]
  >40% | 85
  <=40% | 164
  Not reported/unknown | 2
Left ventricular ejection fraction [Mean (Standard Deviation); unit: %] | 37.5 (16.90)
History of depression [Number; unit: participants]
  Yes | 76
  No | 174
  Unknown/not reported | 1
Geriatric Depression Scale [Mean (Standard Deviation); unit: scores on a scale] — Geriatric Depression Scale (GDS) is a validated self-report measure consisting of 30 questions used to screen elderly people for depression. Cutoff scores are as follows: 0-9 normal, 10-19 mildly depressed, 20-30 severely depressed.
  scores on a scale | 13.3 (3.80)
History of PTSD [Number; unit: participants]
  Yes | 47
  No | 201
  Unknown/not reported | 3
Tobacco use [Number; unit: participants]
  Never smoked | 47
  Former smoker | 154
  Current smoker | 47
  Unknown/not reported | 3
Alcohol use [Number; unit: participants]
  Never | 80
  Former use | 83
  Current use less than or equal to 3 drinks/week | 59
  Current use greater than 3 drinks per week | 29
Marijuana use [Number; unit: participants]
  Never | 156
  Past use | 78
  Current use | 14
  Unknown/not reported | 3
Other illicit substance use [Number; unit: participants]
  Never | 190
  Past use | 57
  Current use | 1
  Unknown/not reported | 3
Received treatment in heart failure specialty clinic [Number; unit: participants]
  Yes | 143
  No | 108
Prescribing providers [Mean (Standard Deviation); unit: prescribing providers] | 5.4 (2.4)
Hospitalizations in past year [Mean (Standard Deviation); unit: hospitalizations] | .58 (1.12)

OUTCOME MEASURES:

1. Primary Outcome: SLUMS Scores
Description: SLUMS (Saint Louis University Mental Status) exam is a validated screening test for cognitive impairment (CI) consisting of 30-point interview scale. SLUMS is considered positive for mild CI if the score is <27 in a person with a high school diploma or <25 in a person who did not complete high school. SLUMS screening is considered positive for severe impairment consistent with dementia if the score is <21 for persons with a high school diploma and <20 for persons who did not complete high school.
Time Frame: baseline collection
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Heart Failure
Number analyzed (Participants) | 251
scores on a scale | 24.39 (4)
Statistical Analysis 1: Comparison: Heart Failure; Descriptive data to describe prevalence of cognitive impairment in outpatient veterans with chronic heart failure; Test type: Superiority or Other; percentage = 57.6

2. Secondary Outcome: Medication Adherence
Description: To capture both overtaking and undertaking medication, a "delta" was determined for each medication by computing the absolute difference between the number of pills taken and the number prescribed over the 30-day period. The delta values for each medication were summed for each individual subject, divided by the total number of pills prescribed, subtracted from 1, and finally multiplied by 100 to obtain an adherence score expressed as a percentage.
Time Frame: 30 days
Measure: Mean (95% Confidence Interval); unit: percentage of adherence
Groups:
- No CI: veteran population with documented heart failure with no cognitive impairment on SLUMS screening test who finished 30-day pill counts
- Mild CI: veteran population with documented heart failure with mild cognitive impairment on SLUMS screening test who finished 30-day pill counts
- Severe CI: veteran population with documented heart failure with severe cognitive impairment (dementia) on SLUMS screening test who finished 30-day pill counts
Arm/Group | No CI | Mild CI | Severe CI
Number analyzed (Participants) | 82 | 66 | 20
percentage of adherence | 81.1 [77.1 to 85.0] | 74.1 [69.6 to 78.5] | 74.0 [65.9 to 82.1]

ADVERSE EVENTS:
Arm/Group | Group 1
Serious Adverse Events (participants affected / at risk) | 0/251
Other Adverse Events (participants affected / at risk) | 0/251

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes